CLINICAL TRIAL: NCT00890565
Title: A Single-Blind, Randomized, Parallel Trial to Define the ECG Effects of Sancuso® (Granisetron Transdermal System) Compared to Placebo and Moxifloxacin in Healthy Men and Women
Brief Title: Safety Study of Electrocardiogram (ECG) Effects of Sancuso® (Granisetron TDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 392MD/39/C
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Electrocardiogram; Effect on electrocardiogram; Granisetron; Moxifloxacin; Pharmacokinetic profile; Sancuso® patch; Transdermal
MeSH Terms: interventions — Granisetron; Sodium Chloride; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A: Sancuso® patch (Experimental): Treatment A: Sancuso® patch (Day 1) and placebo IV (Day 3)
  Interventions: Drug: granisetron
- Treatment B: IV Granisetron 10 mcg/kg (Experimental): Treatment B: placebo patch (Day 1) and granisetron IV (Day 3)
  Interventions: Drug: granisetron
- Treatment C: Matching placebo patch (Placebo Comparator): Treatment C: placebo patch (Day 1) and placebo IV (Day 3)
  Interventions: Drug: granisetron
- Treatment D: Oral Moxifloxacin 400 mg (Active Comparator): Treatment D: placebo patch (Day 1) and oral moxifloxacin (Day 3).
  Interventions: Drug: granisetron

INTERVENTIONS:
Drug: granisetron — Treatment A: Sancuso® patch (3.1mg/24 hours) on Day 1 and IV placebo (0.9% saline) on Day 3 Treatment B: Granisetron IV 10 mcg/kg over 30 seconds on Day 1 and placebo patch on Day 3 Treatment C: Placebo patch on Day 1 and IV placebo on Day 3 Treatment D: 400 mg oral moxifloxacin on Day 1 and placebo patch on Day 3
  Other Names: Granisetron Transdermal System; Sancuso® patch; Kytril®; Granisetron Injection; IV Placebo (0.9% saline); Placebo patches; Avelox® Oral

SUMMARY:
This study aims to evaluate the electrocardiogram (ECG) effects of Sancuso® compared to placebo and moxifloxacin in healthy subjects.

DETAILED DESCRIPTION:
Granisetron is a well tested and established 5-HT3 receptor antagonist used in both oral and intravenous (IV) forms. A transdermal form of granisetron (Sancuso®) was approved by the United States (US) Food and Drug Administration (FDA) in September 2008.

Many of the 5-HT3 antagonists were developed and approved before the adoption of the International Conference on Harmonisation (ICH) E14 standard on QTc and cardiac testing. The association of non-cardiac medicinal products with the potential to prolong the QT interval and induce torsades des pointes (TdP) has significant implications for the future development of medicinal products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* Aged between 18 and 50 years, inclusive, at screening
* BMI between 18.0 and 32.0 kg/m², inclusive

Exclusion Criteria:

* History of drug abuse
* Known hypersensitivity to granisetron, moxifloxacin, or related compounds, such as ciprofloxacin and levofloxacin
* Sustained supine systolic blood pressure >140 mmHg or <100 mmHg or a diastolic blood pressure >95 mmHg at Screening or baseline
* Pulse rate at rest of < 45 bpm or > 100 bpm
* Abnormal Screening ECG indicating a second- or third degree AV block, or one or more of the following: QRS >120 milliseconds (ms); QTcF > 430 (males) or 450 (females) ms; PR interval >240 ms; any rhythm, other than sinus rhythm, interpreted to be clinically significant by the Investigator
* Known history of long-QT syndrome, angina, myocardial ischemia or infarction, congestive heart failure, myocarditis, chest pain or dyspnea on exertion
* Electrolyte disturbances (such as uncorrected hypokalemia/hyperkalemia, hypomagnesemia, hypocalcemia, or hypophosphatemia), idiopathic cardiomyopathy, unexplained syncope, hypertrophic cardiomyopathy, or sudden unexplained death at a young age (< 40 years) in a first-degree relative.
* Has used any medications or consumed any foods contraindicated in the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Time-matched, placebo-corrected change from baseline in QTc based on the Fridericia correction (QTcF). | 0 to 120 hours post-dose

SECONDARY OUTCOMES:
QTc with Bazett correction (QTcB), heart rate, PR interval, QRS interval, uncorrected QT interval, change in ECG morphological patterns and correlation between the QTcF change from baseline and plasma granisetron concentrations | 0 to 120 hours post-dose
Relationship of plasma concentration of granisetron versus QTcF, both graphical and mixed effects analyses of plasma concentration of granisetron versus QTcF will be performed | 0 to 120 hours post-dose
Patch adhesion and residual granisetron after patch use. | 0 to 120 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bridget O'Mahony, PhD, Study Director — Kyowa Kirin Co., Ltd.
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States